CLINICAL TRIAL: NCT02280135
Title: Phase I Clinical Trial of Intravitreal Injection of Autologous Bone Marrow Stem Cells in Patients With Retinitis Pigmentosa
Brief Title: Clinical Trial of Intravitreal Injection of Autologous Bone Marrow Stem Cells in Patients With Retinitis Pigmentosa
Acronym: TC/RP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Spanish National Health System (Other); Hospital Universitario Virgen de la Arrixaca (Other); Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other); Public Health Service, Murcia (Other); Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TC/RP; 2012-000618-12 (EudraCT Number)
Record Dates: First submitted 2014-10-22; First posted 2014-10-31 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravitreal injection of Autologous bone marrow Stem Cell (Experimental): Patients included in the trial will receive a pars plana intravitreal injection of autologous mononuclear cells (MNC) of bone marrow (BM) in one eye (experimental group A or group). The eye in which autologous BM MNCs were injected will be determined randomly.
  The average dose will be 30 million of cells (5-60 million) diluted in 0.1 ml. of saline.
  Interventions: Biological: Intravitreal injection of Autologous bone marrow Stem Cell
- Subconjunctival injection of saline (Placebo Comparator): Patients included in the trial will receive a subconjunctival injection of 0.1 ml of saline (SF) (placebo) in the fellow eye (group B or control group). In this way the patient will receive an injection in the control eye but avoid the risks of intraocular injection.
  Interventions: Other: Subconjunctival injection of saline

INTERVENTIONS:
Biological: Intravitreal injection of Autologous bone marrow Stem Cell — We will proceed to the injection of 0.1 ml of the suspension with the autologous MNC of BM avoiding coincide with conjunctival and scleral hole and perpendicular to the sclera.
  After the injection, a dry, sterile dressing will be placed to prevent reflux. Immediately, the perception of light, the movement of the central retinal artery, the venous pulse and the color of the papilla will be evaluated. If necessary, anterior chamber paracentesis will be performed.
  After injection, the patient will remain with closed eyes and sitting, waiting for cells will be deposited on the bottom of the eyeball and for 3 days will instill tropicamide collyrium every 12 hours.
  Arms: Intravitreal injection of Autologous bone marrow Stem Cell
Other: Subconjunctival injection of saline — In the control eye, will make a subconjunctival injection of 0.1 ml saline. To realize contralateral injection gloves and all surgical materials will change, trying extreme measures of sterility.
  After injection, the patient will remain with closed eyes and sitting, waiting for cells will be deposited on the bottom of the eyeball and for 3 days will instill tropicamide collyrium every 12 hours.
  Arms: Subconjunctival injection of saline

SUMMARY:
The purpose of this study is to evaluate the safety of intravitreal injection of autologous bone marrow stem cells in patients with retinitis pigmentosa by a prospective, single-center, randomized, parallel, double-blind, phase I placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Retinitis Pigmentosa bilateral diagnosis.
* Visual acuity (measured with ETDRS) less than or equal to 20/70 and visual field below 30° central in both eyes.
* Signed informed consent
* Warranty sufficient adherence to protocol. It must fulfill all inclusion criteria.

Exclusion Criteria:

* Concurrence of any systemic or ocular disease that precludes or affects tracking study variables. Specifically retinal involvement with diabetes mellitus, glaucoma, macular degeneration or age.
* Eye surgery in the previous 6 months.
* Patients who are pregnant.
* Patients with active lactation.
* Physically fertile patients, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle or sexual orientation excludes sexual intercourse with a man and women whose partners have been sterilized by vasectomy or other methods, UNLESS tHEY are using a reliable contraceptive method. This birth control method can be:
* Complete abstinence from sexual intercourse
* Surgical sterilization (tubal ligation)
* Surgical sterilization partner (vasectomy)
* Implanted or injectable hormonal contraceptives and oral.
* Patients with cardiac disease, renal, hepatic, systemic, immune that might influence the survival of patients during the test.
* Positive serology for hepatitis B, hepatitis C or HIV.
* Clinical criteria or anesthetics that contraindicate the sedation or the extraction of BM (Altered coagulation system or anticoagulated patient with inability to withdraw anticoagulation, hemodynamic instability, altered skin in the puncture site, etc.)
* Participation in other clinical trials.
* Inability to sign informed consent or understanding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Rate of serious and non-serious adverse events related with the use of bone marrow mononuclear cells in patients with retinitis pigmentosa | 12 months from baseline

SECONDARY OUTCOMES:
Quality of Life: Questionnaire VFQ-25 (Visual Function Questionnaire-25). | 12 months from baseline
Visual acuity (VA): Test ETDRS (Early Treatment Diabetic Retinopathy Study). | 12 months from baseline
Color Vision: Ishihara Color Test. | 12 months from baseline
Contrast sensitivity: CSV-1000E. | 12 months from baseline
Intraocular pressure (IOP): measured in mm Hg with applanation tonometer Haag Streit AT 900. | 12 months from baseline
Examination of the anterior and posterior pole: Made with biomicroscopy (BMC). | 12 months from baseline
Width of retinal macula layer and nerve fiber: Measured with Optical Coherence Tomography Spectral domain (OCT)(Topcon 3D OCT-2000 Spectral Domain OCT). | 12 months from baseline
Visual field (VF) and macular sensitivity (The Humphrey perimeter). | 12 months from baseline
Study eye fundus: Made by Retinography and Angiography fluorescein. | 12 months from baseline
Electrical retinal function: electroretinogram (ERG) (altered / unaltered). | 12 months from baseline
Visual evoked potentials with Pattern Reversal (VEP) (altered / no altered). | 12 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: María Elena Rodriguez González-Herrero, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Clinical Universitary Hospital Virgen de la Arrixaca, El Palmar, Murcia, Spain